CLINICAL TRIAL: NCT00122915
Title: A Prospective, Randomized, Double Blind, Crossover, Multi-center Study to Evaluate the Safety and the Efficacy of Motor Cortex Stimulation With the Cortical Stimulation Lead Model 2976 in Patients With Neuropathic Pain
Brief Title: CONCEPT: Crossover Efficacy Pain Trial in Motor Cortex Stimulation for Intractable Neuropathic Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on a consistently low enrolment rate and procedural challenges that were unknown at study start. It was not based on safety or efficacy concerns.
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CONCEPT
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Pain, Intractable; Facial Pain
Keywords: Motor Cortex Stimulation; Pain treatment; Central post-stroke pain (CPSP); Trigeminal neuropathic pain (TGN); Facial pain; Neurostimuation; Cortical lead; Neuropathic pain
MeSH Terms: conditions — Pain, Intractable; Facial Pain; Agnosia; Neuralgia

INTERVENTIONS:
Device: Cortical lead, 8 electrodes (Model 2976) with Synergy neurostimulator

SUMMARY:
The CONCEPT study has been designed to evaluate the safety and the efficacy of Motor Cortex Stimulation (MCS) with a new cortical lead (circular lead, eight electrodes, Medtronic Inc, Minneapolis, USA) in the treatment of intractable neuropathic pain, in particular for central post-stroke pain (CPSP) and trigeminal neuropathic pain (TGN)/facial pain.

ELIGIBILITY:
Inclusion Criteria:

* CPSP or TGN/facial pain refractory to other medical treatments
* Pain > 1 year prior to baseline
* Pain intensity with an average daily VAS score > 5 demonstrated by 12 ratings across 4 days
* Stable pain medication for > 1 month prior to baseline

Exclusion Criteria:

* CPSP with important paresis/severe motor deficit in the area of pain
* TGN/facial pain with complete deafferentation pain
* Atypical facial pain, i.e. when objective evidence for neuropathic facial pain syndromes is lacking and when specific psychological and behavioral factors can be identified
* Pain associated with malignant neoplastic disease anywhere in the body or head
* History of epilepsy
* Presence of a deterioration of cognitive functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Adverse events reports
Pain assessed by Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Quality of life
Disability
Analgesic, sedative or psychoactive medication intake

CONTACTS AND LOCATIONS:
Overall Officials: Bart Nuttin, PhD, MD, Principal Investigator — UZ Gasthuisberg
Locations (11):
- Universitätsklinik Innsbruck, Universitätsklinik für Neurochirurgie, Innsbruck, Austria
- Belgium (6):
  - Hopital Erasme, Service de Neurochirurgie, Brussels
  - UCL St luc, Neurochirurgie, Brussels
  - AZ St Lucas, Neurochirugie, Ghent
  - UZ Gasthuisberg , Department of Neurosurgery, Leuven
  - CH de la Citadelle, Liège
  - Maria Middelares ZH, Saint Niklaas
- Germany (2):
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Klinikum der Philipps-Universität Marburg, Marburg
- Spain (2):
  - Santa Creu I Sant Pau, Servicio de Neurocirugia, Barcelona
  - Hospital Gregorio Maranon, Servicio de Neurologia, Madrid